CLINICAL TRIAL: NCT01033500
Title: Calcineurin Inhibitor-free, Steroid-free Immunosuppressive Regimen in Simultaneous Islet-Kidney Transplantation for Uremic Type 1 Diabetic Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2010-0042
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Islets of Langerhans Transplantation; Diabetes Mellitus, Type 1; Kidney Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SIK (Experimental): Basiliximab induction with maintenance immunosuppression consisting of belatacept, sirolimus or everolimus, and mycophenolate after simultaneous islet kidney transplantation.
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — Belatacept 10mg/kg on Days 0, 4, 14, 28, 56, and 84 post-transplant, and then 5mg/kg every 4 weeks for the duration of the study.

SUMMARY:
The investigators hypothesize that a calcineurin inhibitor-free, steroid-free, co-stimulatory blockade-based immunosuppressive regimen, in combination with a GLP-1 agonist, will reduce the islet mass required to achieve and sustain insulin independence following simultaneous islet-kidney transplantation.

DETAILED DESCRIPTION:
This is a single center, open-label, non-randomized, prospective, pilot study of 8 Type 1 diabetic/uremic patients, ages 18-60 undergoing simultaneous islet-kidney transplantation. Study to include both male and/or female subjects.

We hypothesize that a calcineurin inhibitor-free, steroid-free, co-stimulatory blockade-based immunosuppressive regimen, in combination with a GLP-1 agonist, will reduce the islet mass required to achieve and sustain insulin independence following simultaneous islet-kidney transplantation.

Furthermore, we anticipate an improvement in creatinine clearance and a reduction in Interstitial Fibrosis/Tubular Atrophy in the transplanted renal allograft, and a reduction of "de novo" human anti-HLA antibody and auto-antibody formation against the respective donors.

Without calcineurin inhibitors or steroids, we hypothesize that belatacept, in conjunction with sirolimus and mycophenolic acid will provide balanced immunosuppression for combined islet-kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include those with Type 1 Diabetes Mellitus, undergoing kidney transplantation, and:

  * are closely followed by a primary care provider and/or endocrinologist for >6 months prior to enrollment in the trial
  * do not have psychogenic factors which preclude therapeutic compliance
  * have a fasting C-peptide of <0.2 ng/mL• have diabetes for >5 years • are between 18 and 65 years of age
  * have a creatinine clearance of less than 20 mL/min
  * have a body mass index of less than or equal to 28
  * In the case of women of childbearing potential (WOCBP), must have a negative pregnancy test and avoid pregnancy throughout the study and 8 weeks after final dose of study drug.
  * WOCBP must use two adequate methods of contraception.
  * A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study and for up to 8 weeks after the last dose of study drug to minimize the risk of pregnancy.

Exclusion Criteria:

* Untreated proliferative diabetic retinopathy

  * HgbA1C >12
  * creatinine clearance > 20 ml/minute
  * presence of panel reactive antibodies (PRA) >20% (per CDC-based assay)
  * malignancy or previous malignancy, except for adequately treated skin cancers (basal cell or squamous cell carcinoma) within the past 5 years
  * sensitivity to iodine and/or shellfish (re: Iothalamate-based GFR testing)
  * x-ray evidence of pulmonary infection
  * active infections
  * active peptic ulcer disease, gall stones, hemangioma, cirrhosis or portal hypertension
  * serological evidence of HIV, HBSAg or HCV
  * abnormal liver function tests (elevated AST and ALT > 2x upper limit of normal)
  * anemia (hemoglobin) <9 gm/dl
  * serum triglycerides >200 mg/dl
  * serum cholesterol >240 mg/dl
  * body mass index above 28
  * unstable cardiovascular status (including positive stress echocardiography if >age 35); severe coexisting cardiac disease, myocardial infarction within the 6 months prior to enrollment in the study, left ventricular ejection fraction of <30%, or evidence of ongoing ischemia
  * prostate specific antigen (PSA) >4 in males >40 years old or with family history of prostate cancer
  * pregnancy or breastfeeding
  * sexually-active females who are not: a) post-menopausal, b) surgically sterile, or c) not using an acceptable method of contraception (oral contraceptives, Norplant, Depo-Provera, and barrier devices are acceptable; condoms used alone are not acceptable)
  * alcohol abuse, substance abuse or smoking within the previous 6 months
  * insulin requirement >1.5 u/kg/day
  * negative for Epstein-Barr virus by IgG determination
  * history of factor V deficiency
  * acute or chronic pancreatitis
  * recurrent attenuated vaccine(s) within the previous 2 months
  * use of an investigational agent within the past 4 weeks
  * sexually active, fertile men not using effective birth control, if their partners are WOCBP
  * prisoners, or subjects who are involuntarily incarcerated
  * subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
  * Previous kidney transplant or previous non-renal transplant
  * kidney transplant from expanded criteria donor (ECD)
  * kidney cold ischemic time projected to be > 20 hours
  * currently receiving immunosuppressive agents for autoimmune disease or other conditions or have comorbidities that treatment with such agents are likely during the trial
  * any condition or circumstance that makes it unsafe to undergo an islet cell or kidney transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Achieve and consistently maintain insulin independence in simultaneous islet-kidney transplant recipients for one year. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fernandez, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States